CLINICAL TRIAL: NCT01736722
Title: Use of MRI-Guided Laser Induced Thermal Therapy (LITT) for Metastatic Brain Tumors
Brief Title: MRI-Guided LITT for Treatment Metastatic Brain Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI change and no enrollment ever, therefore no data available.
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002569
Record Dates: First submitted 2012-11-19; First posted 2012-11-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Brain Tumor
Keywords: Laser Induced Thermal Therapy; Metastatic cancer; Brain Tumor; Visualase; Treatment resistant; Magnetic Resonance Thermal Imaging; Magnetic Imaging
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI-guided laser induced thermal therapy (Experimental): The target tumor/lesion will undergo laser therapy using the MRI scan to plan the treatment and ensure proper placement of the laser within the tumor. An MRI (Magnetic Resonance Imaging) is a exam that creates pictures using magnetic rays instead of x-rays. The tumor(s) will then be heated by the laser in an attempt to eliminate their presence. The physician will be able to see and control the temperature of the laser.
  Interventions: Device: Visualase®

INTERVENTIONS:
Device: Visualase® — The target tumor/lesion will undergo laser therapy using the MRI scan to plan the treatment and ensure proper placement of the laser within the tumor. An MRI (Magnetic Resonance Imaging) is a exam that creates pictures using magnetic rays instead of x-rays. The tumor(s) will then be heated by the laser in an attempt to eliminate their presence. The physician will be able to see and control the temperature of the laser.

SUMMARY:
The Methodist Hospital Neurological Institute is conducting a clinical trial for patients suffering from Metastatic brain tumors. The objective for this study is to evaluate the safety and feasibility of a MRI-guided laser thermal therapy during a real-time MRI guidance for the treatment of brain metastasis.

Patient will undergo laser therapy using the MRI scan to plan the treatment and ensure proper placement of the laser within the tumor. The tumor will then be heated by the laser and monitored by study physicians through the real-time MRI to see and control temperatures in the tissue. One in place, the thermal laser will then surgically remove the lesions. After the procedure, post treatment MR images will thenbe acquired for the determination of the effective treatment region.

DETAILED DESCRIPTION:
This is a study for evaluating the feasibility and safety of MR-guided laser thermal ablation of treatment-resistant brain tumors using the Visualase® Thermal Therapy System (Manufactured by BioTex, Inc., Houston, TX). The Visualase system is FDA cleared for soft tissue ablation in a number of surgical specialties including Neurosurgery (see appendix for documentation). Patients with intracranial brain tumors measuring 3 cm or smaller in largest diameter that have failed any conventional therapy (surgery, stereotactic radiosurgery and/or whole brain radiotherapy) are eligible.

The target tissue containing the tumor will undergo MRI-guided laser induced thermal therapy. MR imaging is used to define the treatment volume as well as plan and verify placement of the applicator. The extent of ablation is quantitatively monitored and displayed during delivery using real-time, MR temperature imaging. MR temperature imaging will also be used to monitor and control the temperature of adjacent tissues. Treatment will be automatically stopped if the MR temperature feedback system reports the temperature in the adjacent tissue has risen above a preset threshold. Treatment can be manually stopped by the neurosurgeon monitoring the treatment in real-time at any point during the procedure by simply turning off the power to the laser from the Visualase® system console. After laser delivery, MR images can be used to verify the extent of treatment and plan a therapy delivery if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. High-grade gliomas, metastatic brain tumors, and other brain tumors refractory to conventional medical therapy.
2. Patient or family able and willing to give informed consent.
3. Subjects with metastatic cancer to the brain who have failed at least one conventional therapy (surgery, stereotactic radio- surgery, chemotherapy, and/or whole brain radiotherapy).
4. Four or fewer previously treated or untreated lesion(s) in the brain.
5. Tumor size ≤ 3.0 cm in largest diameter.
6. MR imaging is not contraindicated for the patient.
7. Lesion(s) are clearly defined on pre-therapy contrast enhanced MRI scans as determined by the treating surgeon.
8. Able and willing to attend all study visits.
9. Karnofsky Performance Scale score >50.
10. Patients age 19 and older.

Exclusion Criteria:

1. Patients or family unwilling or unable to give written consent.
2. Patients who cannot physically fit in, or are too heavy for, the MRI scanner.
3. Patients with contra-indications to MRI imaging, such as, but not limited to, some pacemakers or defibrillators, non- compatible aneurysm clips, shrapnel, or other internal ferromagnetic objects.
4. Known sensitivity to gadolinium-DTPA, or glomerular filtration rate not compatible with receiving gadolinium-DTPA.
5. Based on Treatment Planning Imaging (MR and/or CT):

   * Lesions localized in the brain stem.
   * Lesions less than 5mm from primary branches of cerebral vessels, venous sinus, hypophysis or cranial nerves.
   * Presence of more than 4 brain tumors at the time of enrollment.
   * Medical issues which prohibit the patient from undergoing surgery (as determined by the treating surgeon, anesthesiologist, IMPAC clinic, referring physician).
   * Positive pregnancy test for women of child-bearing age.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2014-03-05 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility | 30d
  Safety: To determine that the procedure can be safely tolerated without adverse events based on day 30 procedure-related morbidity and mortality. Feasibility: To determine that the the rate of technical success or failure to complete the initial procedure with no associated major complications.

SECONDARY OUTCOMES:
Number of patients with survival | 30 days
  30 day imaging evaluation of the laser induced lesion Correlation: examination of the extent to which Visulase predictions based on MRTI data match lesion dimensions from post-therapy MRI assessments. Estimates of durations, required facilities, required personnel, and costs for all aspects of the treatment procedure. Local control of lesions at 30 day as defined by volume of lesion increasing by no more than 25%.
  Accrual of patient survival post Visualase therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Z New, M.D., Principal Investigator — Methodist Neurological Institute
Locations (1):
- Methodist Neurological Institute - Department of Neurosurgery, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this time.

REFERENCES:
- See also: Related Info — http://www.methodisthealth.com/ni.cfm?id=35605